CLINICAL TRIAL: NCT07114107
Title: Evaluation of the Efficacy and Safety of Vibroacoustic Therapy With Oscillating Positive Expiratory Pressure in the Treatment of Nasal Congestion: A Randomized, Double-Blind, Placebo-Controlled Parallel-Group Clinical Trial
Brief Title: Vibroacoustic Therapy With Oscillating Positive Expiratory Pressure in the Treatment of Nasal Congestion
Acronym: VAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Huzhou Central Hospital (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-0820
Record Dates: First submitted 2025-07-16; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-05

CONDITIONS: Atopic Rhinitis; Atopic Asthma
Keywords: nasal congestion; Vibroacoustic therapy; Oscillating Positive Expiratory Pressure
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Nasal Obstruction | interventions — Histamine Antagonists

STUDY DESIGN:
Intervention Model Description: A Randomized, double-Blind, Multi-Center，Placebo-Controlled Parallel-Group Clinical Trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- treatment group 1-nasal congestion with only atopic rhinitis (Experimental): this group participants use the acoustic vibration device therapy device, respectively, 3 times a day for 3 minutes each time for 2 month
  Interventions: Device: VPAT (Vibratory Positive Pressure Therapeutic Apparatus）; Drug: basic medications (antihistamines, mometasone furoate nasal spray, ICS-LABA
- treatment group 2-nasal congestion with atopic rhinitis and atopic asthma (Experimental): this group participants use the acoustic vibration device therapy device, respectively, 3 times a day for 3 minutes each time for 2 month
  Interventions: Device: VPAT (Vibratory Positive Pressure Therapeutic Apparatus）; Drug: basic medications (antihistamines, mometasone furoate nasal spray, ICS-LABA
- control group 1-nasal congestion with only atopic rhinitis (Active Comparator): this group participants use the oscillating positive expiratory pressure therapy device (without acoustic function), respectively, 3 times a day for 3 minutes each time for 2 months.
  Interventions: Drug: basic medications (antihistamines, mometasone furoate nasal spray, ICS-LABA; Device: OPEP（Oscillating Positive Expiratory Pressure device）
- control group 2-nasal congestion with atopic rhinitis and atopic ashtma (Active Comparator): this group participants use the oscillating positive expiratory pressure therapy device (without acoustic function), respectively, 3 times a day for 3 minutes each time for 2 months.
  Interventions: Drug: basic medications (antihistamines, mometasone furoate nasal spray, ICS-LABA; Device: OPEP（Oscillating Positive Expiratory Pressure device）

INTERVENTIONS:
Device: VPAT (Vibratory Positive Pressure Therapeutic Apparatus） — VPAT (Vibratory Positive Pressure Therapeutic Apparatus）is a physical solution which can relieve nasal congestion and discomforts by applying acoustic vibration and oscillatory positive expiratory pressure. Clinical research has shown that low-frequency vibration at approximately 130 Hz promotes the production of the highest concentration of Nitric Oxide (NO) in the paranal sinuses, which helps to regulate the nasal mucosal blood, restoring the mucous membrance-cilia mechanism, clean up the bacteria, viruses and allergenic particles in the respiratory tract.
  Combined with Oscillatory Positive Expiratory Pressure and Transnasal Breathing, it can help to cultivate the habit of nasal breathing and slow breathing, as well as to restore the function of lungs.
  Arms: treatment group 1-nasal congestion with only atopic rhinitis; treatment group 2-nasal congestion with atopic rhinitis and atopic asthma
Drug: basic medications (antihistamines, mometasone furoate nasal spray, ICS-LABA — All participants need basic control drugs contains antihistamines(Ebastine 10 mg once daily for 2 weeks), mometasone furoate nasal spray(Spray 2 puffs into each nostril, each puff contains 50 μg of mometasone furoate, i.e., 100 μg per administration, once daily for 2 weeks).
  Asthma participants should added Inhaled corticosteroids-long-acting beta-agonists (ICS-LABA) therapy. For mild to moderate asthma: budesonide/formoterol (160μg/4.5μg) , with 1 inhalation each time, twice daily, or salmeterol/fluticasone propionate (50μg/100μg) with 1 inhalation each time, twice daily. For moderate to severe asthma: Budesonide/Formoterol (320μg/4.5μg), with 1 inhalation each time, twice daily; or salmeterol/fluticasone propionate (50μg/250μg or 50μg/500μg) with 1 inhalation each time, twice daily. Dosage adjustments should be evaluated and determined by the physician based on the patient's disease control status.
Device: OPEP（Oscillating Positive Expiratory Pressure device） — Oscillating Positive Expiratory Pressure (OPEP) device contain a inner ball that creates a resistance and oscillates when the patient blows through the device. This resistance helps splint the airways open during exhalation whilst the oscillation loosens the mucous within the airways. This makes it easier for some patients to clear their sputum.
  Arms: control group 1-nasal congestion with only atopic rhinitis; control group 2-nasal congestion with atopic rhinitis and atopic ashtma

SUMMARY:
This is a prospective study. It enrolls subjects with allergic rhinitis, with or without asthma, who have nasal congestion as the main symptom and meet the inclusion criteria, aiming to evaluate the efficacy and safety of acoustic vibration combined with an oscillating positive expiratory pressure device in the treatment of patients with nasal congestion. On the premise that subjects agree to use basic medications (antihistamines, mometasone furoate nasal spray, ICS-LABA), they are instructed to use the acoustic vibration therapy device and the oscillating positive expiratory pressure therapy device respectively, 3 times a day for 3 minutes each time. Indicators related to nasal congestion will be measured immediately after a single use, as well as at 2 weeks, 4 weeks, and 8 weeks of use, so as to monitor the improvement of nasal ventilation and accompanying symptoms in the subjects.

DETAILED DESCRIPTION:
Objective: To evaluate the efficacy and safety of acoustic vibration combined with an oscillating positive expiratory pressure device in the treatment of patients with nasal congestion.

Methods: A total of 200 subjects with nasal congestion as the main symptom who met the inclusion criteria were enrolled in this study. Among them, 100 subjects were treated with an acoustic vibration therapy device (treatment group), including 50 subjects with allergic rhinitis and 50 subjects with allergic rhinitis complicated with asthma; the other 100 subjects were treated with an oscillating positive expiratory pressure therapy device (without acoustic function, only with oscillating positive expiratory pressure function) as the control group, which also included 50 subjects with allergic rhinitis and 50 subjects with allergic rhinitis complicated with asthma. On the premise that subjects agreed to use basic medications (antihistamines, mometasone furoate nasal spray, ICS-LABA), they were instructed to use the acoustic vibration therapy device or the oscillating positive expiratory pressure therapy device, respectively, 3 times a day for 3 minutes each time. Nasal congestion-related indicators were measured immediately after a single use, as well as at 2 weeks, 4 weeks, and 8 weeks of use. The improvement of nasal ventilation and accompanying symptoms was monitored to clarify the efficacy and safety of the two devices.

Key Inclusion Criteria:

Subjects aged 12-50 years at the time of signing the informed consent form, regardless of gender;Meeting the guideline diagnostic criteria for allergic rhinitis with or without asthma;Presenting with significant nasal congestion for at least 1 week, with or without asthma, and symptoms poorly controlled despite the use of intranasal glucocorticoids and/or other therapeutic drugs;Patients with moderate to severe seasonal allergic rhinitis (SAR) with a mean Total Nasal Symptom Score (TNSS) ≥ 9 points, including nasal congestion ≥ 3 points;Willing and able to complete follow-up visits and scoring assessments at 2 weeks, 4 weeks, and 8 weeks during the study period as required by the protocol;Regular use of standard medications;Willing to receive treatment with acoustic vibration or oscillating positive expiratory pressure device 3 times a day for 3 minutes each time, and perform corresponding check-in and reporting;Voluntarily signing the informed consent form before the start of any study-related procedures, able to communicate smoothly with researchers, understand and be willing to strictly comply with the requirements of this clinical study protocol to complete the study.

Expected Outcomes:

Statistically significant improvements in relevant parameters in the oscillating positive expiratory pressure therapy device group after treatment, including: Peak Nasal Inspiratory Flow (PNIF), Peak Expiratory Flow (PEF), Fractional Exhaled Nitric Oxide(FeNO), Visual Analogue Scale (VAS), Total Nasal Symptom Score + Total Non-Nasal Symptom Score (TNSS + TNNSS), Rhinitis-Related Quality of Life Questionnaire (RQLQ), Asthma Control Test (ACT), Asthma Quality of Life Questionnaire (AQLQ), anterior rhinoscope (ENT), Pulmonary Function Tests, etc. The safety of acoustic vibration therapy device and oscillating positive expiratory pressure therapy device in the treatment of nasal congestion will be clarified, specifically including the incidence of adverse events such as no epistaxis, dyspnea, etc.

Hypothesis:

In the treatment of subjects with nasal congestion as the main symptom, whether they have simple allergic rhinitis or allergic rhinitis complicated with asthma, nasal congestion and related symptoms are significantly improved after daily treatment with acoustic vibration or oscillating positive expiratory pressure devices 3 times a day.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 12-50 years at the time of signing the informed consent form, regardless of gender; Meeting the guideline diagnostic criteria for allergic rhinitis with or without asthma; Presenting with significant nasal congestion for at least 1 week, with or without asthma, and symptoms poorly controlled despite the use of intranasal glucocorticoids and/or other therapeutic drugs; Patients with moderate to severe seasonal allergic rhinitis (SAR) with a mean Total Nasal Symptom Score (TNSS) ≥ 9 points, including nasal congestion ≥ 3 points; Willing and able to complete follow-up visits and scoring assessments at 2 weeks, 4 weeks, and 8 weeks during the study period as required by the protocol; Regular use of standard medications; Willing to receive treatment with acoustic vibration or oscillating positive expiratory pressure device 3 times a day for 3 minutes each time, and perform corresponding check-in and reporting; Voluntarily signing the informed consent form before the start of any study-related procedures, able to communicate smoothly with researchers, understand and be willing to strictly comply with the requirements of this clinical study protocol to complete the study.

Exclusion Criteria:

* Exclusion criteria identified by pre-examination with nasal endoscopy include: definite structural/mechanical obstruction (moderate-to-severe nasal septum deviation, moderate-to-severe nasal valve collapse, grade 3-4 nasal polyps, and inferior turbinate hypertrophy that may reduce decongestion reversibility); A history of severe epistaxis within 3 months, or use of anticoagulants; Complicated with unstable asthma; Patients currently receiving special treatment regimens, including biologic therapy and dust mite desensitization therapy; Complicated with major diseases of the respiratory or cardiovascular system: such as moderate-to-severe COPD, coronary heart disease, bronchiectasis, pulmonary infection, or respiratory tract infection; Suffering from malignant tumors or having a history of malignant tumors (except for cutaneous squamous cell carcinoma, basal cell carcinoma, or cervical carcinoma in situ that have been completely resected with no evidence of recurrence); Having undergone major surgery within 3 months before randomization, or planning to undergo major surgery during the study period; Suffering from severe concomitant diseases or other conditions that, in the investigator's judgment, make the patient unsuitable for participation in this trial.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Peak Nasal Inspiratory Flow (PNIF) | These indicators are measured at baseline, immediately after a single use, and at 2 weeks, 4 weeks, and 8 weeks of use.
  PNIF is a simple, portable inspiratory flow meter, which measures PNIF (peak nasal inspiratory flow) through the nasal passage; providing information of nasal obstruction. Objective measurement of nasal obstruction is useful in the diagnosis of a number of conditions and establishing efficacy of nasal decongestants, it can be Individually calibrated and used during assessment of allergic rhinitis.

SECONDARY OUTCOMES:
Peak Expiratory Flow (PEF) | These indicators are measured at baseline, immediately after a single use, and at 2 weeks, 4 weeks, and 8 weeks of use.
VAS (Visual Analogue Scale ) | These indicators are measured at baseline, immediately after a single use, and at 2 weeks, 4 weeks, and 8 weeks of use.
Total Nasal Symptom Score + Total Non-Nasal Symptom Score (TNSS + TNNSS) | These indicators are measured at baseline, 2 weeks, 4 weeks, and 8 weeks of use.
RQLQ(Rhinitis-Related Quality of Life Questionnaire ) | These indicators are measured at baseline, 2 weeks, 4 weeks, and 8 weeks of use.
FeNO (Fractional Exhaled Nitric Oxide) | These indicators are measured at baseline, immediately after a single use, and at 2 weeks, 4 weeks, and 8 weeks of use.
ACT(Asthma Control Test ) | These indicators are measured at baseline, 2 weeks, 4 weeks, and 8 weeks of use.
AQLQ(Asthma Quality of Life Questionnaire ) | These indicators are measured at baseline, 2 weeks, 4 weeks, and 8 weeks of use.
anterior rhinoscope | These indicators are measured at baseline, 2 weeks, 4 weeks, and 8 weeks of use.The anterior rhinoscope is used to examine for the presence of bleeding, aggravated ulcers.
  The anterior rhinoscope is used to examine for the presence of bleeding, aggravated ulcers, and other conditions, so as to ensure that adverse reactions such as increased bleeding and severe hemorrhage (which may result from the potential aggravation of ulceration and erosion in areas like the nasal vestibule) do not occur during the treatment process.
Pulmonary Function Test FEV1/FVC ratio | up to 8 weeks
  We will examine the patients' pulmonary function test data at the time of enrollment and after 8 weeks of treatment, respectively. Specifically, this will mainly include improvements in the statistical results of FEV1/FVC%Pred (predicted percentage of forced expiratory volume in 1 second to forced vital capacity ratio)
Pulmonary Function Test | up to 8 weeks
  We will examine the patients' pulmonary function test FEV1%Pred (predicted percentage of forced expiratory volume in 1 second).

CONTACTS AND LOCATIONS:
Overall Officials: Huiying Wang, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Huiying Wang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes